CLINICAL TRIAL: NCT05479370
Title: Investigation and Comparison of the Antibody Response Initiated by Recombinant, Cell-Based and Egg-Based Influenza Vaccines
Brief Title: Immunogenicity Trial of 3 Influenza Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: A*Star (Other); University of Melbourne (Other); Sanofi (Industry)
Responsible Party: Principal Investigator, Barnaby Young, Principal Investigator, Head of Singapore Infectious Disease Clinical Research Network, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022/00275
Record Dates: First submitted 2022-07-12; First posted 2022-07-29 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2024-10

CONDITIONS: Influenza Vaccination
Keywords: Humoral immunity; Antibody; Vaccination history; B cell response; Vaccine efficacy
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Frequently vaccinated Group 1: QIV-R (Experimental): Frequently vaccinated participants (3 or more influenza vaccinations during the preceding 5 years) received a 0.5mL dose of Flublok Quadrivalent vaccine, intra-muscularly, at Day 0.
  Interventions: Biological: Flublok Quadrivalent vaccine
- Frequently vaccinated Group 2: QIV-E (Experimental): Frequently vaccinated participants (3 or more influenza vaccinations during the preceding 5 years) received a 0.5mL dose of Fluarix Quadrivalent vaccine, intra-muscularly, at Day 0.
  Interventions: Biological: Fluarix Quadrivalent vaccine
- Frequently vaccinated Group 3: QIV-C (Experimental): Frequently vaccinated participants (3 or more influenza vaccinations during the preceding 5 years) received a 0.5mL dose of Flucelvax Quadrivalent vaccine, intra-muscularly, at Day 0.
  Interventions: Biological: Flucelvax Quadrivalent vaccine
- Infrequently vaccinated Group 4: QIV-R (Experimental): Infrequently vaccinated participants (0 or 1 influenza vaccination during the preceding 5 years) received a 0.5mL dose of Flublok Quadrivalent vaccine, intra-muscularly, at Day 0.
  Interventions: Biological: Flublok Quadrivalent vaccine
- Infrequently vaccinated Group 5: QIV-E (Experimental): Infrequently vaccinated participants (0 or 1 influenza vaccination during the preceding 5 years) received a 0.5mL dose of Fluarix Quadrivalent vaccine, intra-muscularly, at Day 0.
  Interventions: Biological: Fluarix Quadrivalent vaccine
- Infrequently vaccinated Group 6: QIV-C (Experimental): Infrequently vaccinated participants (0 or 1 influenza vaccination during the preceding 5 years) received a 0.5mL dose of Flucelvax Quadrivalent vaccine, intra-muscularly, at Day 0.
  Interventions: Biological: Flucelvax Quadrivalent vaccine

INTERVENTIONS:
Biological: Flublok Quadrivalent vaccine — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Arms: Frequently vaccinated Group 1: QIV-R; Infrequently vaccinated Group 4: QIV-R
Biological: Fluarix Quadrivalent vaccine — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Arms: Frequently vaccinated Group 2: QIV-E; Infrequently vaccinated Group 5: QIV-E
Biological: Flucelvax Quadrivalent vaccine — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Arms: Frequently vaccinated Group 3: QIV-C; Infrequently vaccinated Group 6: QIV-C

SUMMARY:
This study is a prospective randomised trial of 3 influenza vaccine formulations with different manufacturing processes: 1) egg-grown (QIV-E); 2) cell-grown (QIV-C); and 3) recombinant protein (QIV-R). The main objective is to compare the antibody responses following influenza vaccination among these 3 vaccines to determine whether recombinant vaccines offer superior protection over standard egg or cell-based formulations. The attenuating effects of prior vaccination on vaccine immunogenicity will also be evaluated.

Hypothesis: Vaccination with recombinant vaccine results in better antibody responses, particularly against A(H3N2) viruses, than either standard egg-grown vaccines or cell-grown vaccines.

DETAILED DESCRIPTION:
Influenza vaccine effectiveness varies from year to year and is generally poorest against A(H3N2), the virus subtype for which genetic and antigenic evolution among circulating strains has been greatest. While vaccination may stimulate robust antibody responses to vaccine antigen, the breadth of antibodies generated may be insufficient to protect vaccinees from infection by all circulating viruses. Furthermore, vaccine-induced antibody responses may become blunted after repeated vaccinations. However, investigations to-date have largely only examined antibody titres against the vaccine antigen, and have mostly not considered vaccination history.

In recent years, problems associated with egg-based production of vaccine strains have exacerbated these problems. Influenza viruses generally acquire substitutions within the hemagglutinin (HA) protein to adapt to growth in eggs. In the case of A(H3N2) viruses these adaptations often render them antigenically distinct from the wildtype virus. Subsequently, antibodies induced against egg-adapted epitopes in the vaccine will provide limited protection against infection by circulating viruses, and vaccine effectiveness has been very low. Cell-based vaccines have been developed which can overcome some of the problems associated with egg manufacturing, but both egg and cell-based vaccines depend on the growth and purification of live viruses that must be inactivated and split before being formulated into vaccines. The chemical inactivation process disrupts key antigenic structures and alters vaccines' antigenicity, and are thus likely to impact vaccine efficacy. The Sanofi recombinant vaccine Flublok® uses a recombinant technology to produce purified HA in an un-cleaved form that is unable to mediate endosomal and viral membrane fusion. Importantly the manufacturing process does not require any chemical inactivation, meaning that the HA proteins are not exposed to any potential cross-linking agents that may alter antigenicity of the vaccine. In addition, Flublok® contains a higher concentration of antigen than standard-dose vaccines with 45 μg of each antigen included. A recent comparative analysis of antibody response from healthy adults (18-49 years old), comparing egg-based, cell-based and recombinant (Flublok®) vaccines found that Flublok® resulted in significantly higher titres of neutralizing antibody and that the recombinant vaccine may have properties that allow for better viral neutralisation compared to traditional cell-based vaccines. As such, clinical efficacy gains could be associated with differences between the HA in the different vaccines.

This study will assess the immunogenicity of QIV-R (Flublok) against QIV-E (Fluarix) and QIV-C (Flucelvax) vaccines, and investigate the attenuating effects of prior vaccination on vaccine immunogenicity. It will be a randomized, modified double-blind study conducted in Singapore on 360 adults, aged 21-49 years. Randomisation will be stratified by vaccination history, frequently vaccinated (3+ vaccinations during the preceding 5 years) vs. infrequently vaccinated (0-1 vaccination during the preceding 5 years), to compare the responses to each vaccine. This study is powered to primarily assess the immunogenicity (as assessed by haemagglutination inhibition (HI) geometric mean titres (GMTs) at 14-21 days post-vaccination) of QIV-R compared with QIV-E and QIV-C. Pre-vaccination, post-vaccination and post-season serum samples will be tested for antibody titres against the 4 vaccine strains in QIV-R, QIV-C and QIV-E vaccines via HI assays. For some A(H3N2) and B viruses, a microneutralisation (MN) assay will be used to assess the ability of antibodies to neutralize virus infectivity. Over the 1 year follow up period, participants who report acute respiratory infection (ARI) symptoms will have their respiratory swabs collected and tested for Influenza using reverse transcription real-time polymerase chain reaction (RT-PCR). Influenza-positive samples will be forwarded to the WHOCCRRI for virus characterization. The virus subtype (for influenza A) or lineage (for influenza B) will be identified. Viruses will be isolated and tested by HI/MN or similar assay to assess antigenic match to vaccine, and sequenced to assess genetic match to the vaccine and to identify any genetic clusters. Peripheral blood mononuclear cells (PBMCs) will be stained with up to four fluorescent labelled recombinant HA probes representing the vaccine strain and prior A(H3N2) vaccine strains, together with monoclonal antibodies against B cell activation and differentiation markers and isotypes (IgG, IgG3, IgM, IgA, IgD) to compare the magnitude of total HA-reactive B cell response and HA cross-reactivity profiles.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Willing and able to provide 4 blood samples at D0, 14, 150 and 330 post-vaccination
* Has not received influenza vaccine for at least 6 months
* Willing to provide current mobile phone number for SMS reminders

Exclusion Criteria:

* Known contraindication(s) for QIV (e.g. hypersensitivity to vaccine component (including eggs)).
* Recently (last 7 days) or currently ill or has a fever above 38 degrees celsius
* Cannot recall if they were vaccinated against influenza during more or less than two of the preceding five years. Vaccinated during two of the preceding five years.
* Hypogammaglobulinaemia on immunoglobulin replacement
* Undergoing immunosuppressive therapies including corticosteroids

Ages: 21 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 366 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Antibody titres against the 4 vaccine antigens | Day 0, 14, 150, 330
  Post-vaccination geometric mean titre in each vaccination group as measured by the haemagglutination inhibition assay, adjusted for vaccination history and baseline titre.

SECONDARY OUTCOMES:
Pre- to post-vaccination antibody titre ratio between vaccination groups | Day 0, 14, 150, 330
  Pre- to post-vaccination mean fold rise in geometric mean antibody titre between QIV-R, QIV-C and QIV-E.
Range of influenza A(H3N2) strains recognized by the antibodies | Day 0, 14, 150, 330
  Breadth of antibodies induced by vaccination as measured through pre-vaccination, post-vaccination and post-season serum samples tested against a landscape panel of approximately 30 influenza A(H3N2) strains that have circulated since 1968.
Attenuating effects of prior vaccination on antibody titres | Day 0, 14, 150, 330
  For each vaccine type and vaccination history group (frequently versus infrequently vaccinated), post-vaccination geometric mean titre will be compared.
Attenuating effects of prior vaccination on vaccine immunogenicity | Day 0, 14, 150, 330
  For each vaccine type and vaccination history group (frequently versus infrequently vaccinated), antibody breadth (proportion of landscape antigens with geometric mean titre>40) will be compared.
Long-term humoral immunity | Day 0, 14, 150, 330
  Antibody titres against vaccine antigens up to 12 months after vaccination will be compared between vaccination groups using post-season geometric mean titre.
Long-term vaccine immunogenicity | Day 0, 14, 150, 330
  Antibody titres against vaccine antigens up to 12 months after vaccination will be compared between vaccination groups using proportion of landscape antigens with geometric mean titre>40.
B cell responses | Day 0, 14, 150, 330
  Heterogeneity of antibody generating B cells in terms of phenotype and reactivity against a panel of well-defined recombinant hemagglutinin probes that represent a range of influenza A(H3N2) virus clades will be measured.
Vaccine efficacy | Day 0, 14, 150, 330
  Proportion of participants who are infected with Influenza virus within the 1 year study period will be assessed.
Antibody titres in influenza virus-infected versus uninfected participants | Day 0, 14, 150, 330
  Post-vaccination geometric mean titre in infected versus uninfected participants for each vaccination group will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Barnaby Young, Dr, Principal Investigator — National Centre for Infectious Diseases
Locations (1):
- National Centre for Infectious Diseases (NCID), Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data and data dictionary
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After study publication.
Access Criteria: All researchers.

REFERENCES:
- [Background] Gouma S, Zost SJ, Parkhouse K, Branche A, Topham DJ, Cobey S, Hensley SE. Comparison of Human H3N2 Antibody Responses Elicited by Egg-Based, Cell-Based, and Recombinant Protein-Based Influenza Vaccines During the 2017-2018 Season. Clin Infect Dis. 2020 Sep 12;71(6):1447-1453. doi: 10.1093/cid/ciz996. PMID 31598646
- [Background] Wang W, Alvarado-Facundo E, Vassell R, Collins L, Colombo RE, Ganesan A, Geaney C, Hrncir D, Lalani T, Markelz AE, Maves RC, McClenathan B, Mende K, Richard SA, Schofield C, Seshadri S, Spooner C, Utz GC, Warkentien TE, Levine M, Coles CL, Burgess TH, Eichelberger M, Weiss CD. Comparison of A(H3N2) Neutralizing Antibody Responses Elicited by 2018-2019 Season Quadrivalent Influenza Vaccines Derived from Eggs, Cells, and Recombinant Hemagglutinin. Clin Infect Dis. 2021 Dec 6;73(11):e4312-e4320. doi: 10.1093/cid/ciaa1352. PMID 32898271

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT05479370/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT05479370/ICF_001.pdf